CLINICAL TRIAL: NCT05797519
Title: Clinical Safety and Efficacy of the VDyne Transcatheter Tricuspid Valve Replacement System for the Treatment of Tricuspid Regurgitation
Acronym: VISTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VDyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR0038-P
Record Dates: First submitted 2023-03-06; First posted 2023-04-04 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Disease; Tricuspid Valvular Disorders
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- VDyne System Treatment Arm (Experimental)
  Interventions: Device: VDyne Transcatheter Tricuspid Valve Replacement System

INTERVENTIONS:
Device: VDyne Transcatheter Tricuspid Valve Replacement System — The study investigational device is the VDyne Transcatheter Tricuspid Valve Replacement System.
  Other Names: VDyne System; VDyne Tricuspid System; VDyne Valve System; VDyne Valve

SUMMARY:
The purpose of this clinical study is to collect safety and efficacy data of the VDyne System to support Conformitè Europëenne (CE) Mark of the VDyne System.

ELIGIBILITY:
Inclusion Criteria:

1. Severe or greater tricuspid valve regurgitation of primary or secondary etiology.
2. NYHA class ≥ II. If NYHA Class IV, patient must be ambulatory.
3. Subject is adequately treated with medical therapy for heart failure >30 days prior to index procedure, including a diuretic.
4. Heart Team determines patient is a recommended candidate for the VDyne System.
5. Age 18 years or older at time of the index procedure.
6. Clinical Screening Committee (CSC) and Imaging Core Labs confirm suitability for treatment with the VDyne System.

Exclusion Criteria:

VDYNE SYSTEM SUITABILITY

1. Patient anatomy (cardiac and vascular) is not suitable for the VDyne System as assessed by Imaging Core Labs, Sponsor and/or Clinical Screening Committee (CSC)
2. Intolerance to procedural anticoagulation or post-procedural antiplatelet/anticoagulation regimen that cannot be medically managed
3. Hypersensitivity to nickel or titanium

   CLINICAL EXCLUSION CRITERIA (assessed by pre-procedural imaging)
4. Left Ventricular Ejection Fraction (LVEF) <30%
5. Severe RV dysfunction as assessed by the Clinical Screening Committee (CSC).
6. Significant abnormalities of the tricuspid valve and sub-valvular apparatus
7. Sepsis including active infective endocarditis (IE) (within the last 6 months)
8. Right ventricular, atrial thrombus, vegetation or mass on tricuspid valve.
9. Severe tricuspid annular or leaflets calcification
10. Systolic pulmonary hypertension with systolic pulmonary artery pressure >70 mmHg or pulmonary vascular resistance (PVR) >5 wood units as determined by RHC.
11. History of rheumatic fever that impacts the native tricuspid valve or surrounding structures.

    CONCOMITANT PROCEDURES
12. Significant coronary artery disease requiring treatment such as symptomatic, unresolved multi-vessel or unprotected left main coronary artery disease (CAD).
13. Any planned surgery or interventional procedure within 30 days prior to or following the implant procedure. This includes any planned concomitant cardiovascular procedure [e.g. Coronary Artery Bypass Grafting (CABG), percutaneous coronary intervention (PCI), pulmonary vein ablation, left atrial appendage occlusion, septal defect repair, etc.]
14. Unresolved severe symptomatic carotid stenosis (> 70% by ultrasound)
15. Cardiac resynchronization therapy device or implantable pulse generator implanted within 60 days of planned implant procedure.
16. Permanent pacing leads that will interfere with delivery or implantation of the VDyne Valve.
17. Cardiogenic shock or hemodynamic instability requiring inotropes or mechanical support devices at the time of planned implant procedure.
18. Prior tricuspid valve surgery or catheter-based therapy with permanent residual device(s) implanted that would preclude delivery or implantation of the VDyne Valve (e.g. valve replacement, edge to edge repair, etc.)
19. Significant valvular heart disease requiring intervention other than the tricuspid valve
20. Known significant intracardiac shunt [e.g. septal defect), patent foramen ovales (PFOs) without significant shunts are allowed]

    COMORBIDITIES
21. Cerebrovascular accident (stroke, TIA) within 6 months of treatment procedure
22. Severe lung disease [severe chronic obstructive pulmonary disease (COPD) or continuous use of home oxygen or oral steroids]
23. Acute myocardial infarction (AMI) within 30 days
24. Significant renal dysfunction (eGFR<30 ml/min/1.73m2) or on dialysis
25. End-stage liver disease (MELD > 11 and Child-Pugh class C)
26. Bleeding requiring transfusion within 30 days
27. Coagulopathy or other clotting disorder that cannot be medically managed
28. Chronic immunosuppression or other condition that could impair healing response
29. Any of the following: leukopenia, chronic anemia [Hemoglobin (Hgb) < 9], current thrombocytopenia (platelets <70), history of bleeding diathesis, or coagulopathy
30. Unwilling to receive blood products GENERAL EXCLUSION CRITERIA
31. Known hypersensitivity or contraindication to procedural or post-procedural medications (e.g., contrast solution) which cannot be adequately managed medically
32. Life expectancy less than 12 months due to non-cardiac comorbidities
33. Treatment is not expected to provide benefit (futile)
34. Current IV Drug user (must be free drug abuse for > 1 year)
35. Pregnant, lactating or planning pregnancy during the course of the study
36. Vulnerable patient groups (minors, cognitively impaired persons, prisoners, persons whose willingness to volunteer could be unduly influenced by the expectation of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate, such as students, residents, and employees)
37. Currently participating in an investigational drug or device trial that has not reached its primary endpoint or is likely to interfere with this study
38. Patient (or legal guardian) unable or unwilling to provide written informed consent before study-specific procedures are conducted
39. Patient unable or unwilling to comply with study required testing and follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) | 30 days post-procedure
  The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) within 30 days of the procedure, as classified by the Clinical Events Committee (CEC).
Change in tricuspid valve regurgitation as measured by the Imaging Core Labs | From Baseline to 1 month post-procedure
  Change in tricuspid valve regurgitation as measured by the Imaging Core Labs
Changes in quality of life as measured by the KCCQ changes. | From Baseline to 1 month post-procedure
  Changes in quality of life as measured by the KCCQ changes. Higher score indicates worse outcome.
Changes in functional capacity (6-minute walk test) | From Baseline to 1 month post-procedure
  Changes in functional capacity (6-minute walk test)
Changes in symptom status (NYHA class) | From Baseline to 1 month post-procedure
  Changes in symptom status (NYHA class)

SECONDARY OUTCOMES:
The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) | From Baseline to 1 year post-procedure
  The percentage of subjects with Device- and/or Procedure related Major Adverse Events as classified by the CEC
Change in tricuspid valve regurgitation as measured by the Imaging Core Lab | From Baseline to 3 months, 6 months and 1 year
  Change in tricuspid valve regurgitation as measured by the Imaging Core Lab
Intra-Procedural success | From implant start time to procedure room exit
  Rate of successful implantation of the VDyne Valve using the VDyne Delivery System, absence of procedural mortality or stroke, adequate performance of the VDyne Valve, no device-related obstruction of forward flow or pulmonary embolism and & freedom from emergency surgery or reintervention during the first 24 hours related to the device or access procedure.
Clinical success | From implant to 30 days post implant
  Absence of procedural mortality, proper position of the device with adequate performance, freedom from unplanned surgical or interventional procedures related to the device or procedure, absence of major adverse events, device related pulmonary embolism and obstruction of forward flow, any severe hemodynamic compromise leading to heart transplantation or major cardiac assistance or any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention.
Changes in symptom status (NYHA class) | From Baseline to 3 months, 6 months and 1 year
  Changes in symptom status (NYHA class)
Changes in functional capacity (6 minute walk test) | From Baseline to 3 months, 6 months and 1 year
  Changes in functional capacity (6 minute walk test)
Changes in quality of life as measured by the KCCQ changes. | From Baseline to 3 months, 6 months and 1 year
  Changes in quality of life as measured by the KCCQ changes. Higher score indicates worse outcome.
Clinical success | From implant to 1 Year post-implant
  No rehospitalizations or reinterventions for the underlying condition (e.g., tricuspid regurgitation/stenosis, heart failure);
Clinical success | From implant to 1 Year post-implant
  Improvement from baseline in symptoms (e.g., NYHA improvement by >1 functional class); and/or Improvement from baseline in functional status (e.g., 6-min walk test improvement by >30 m); and/or Improvement from baseline in quality-of-life (e.g., Kansas City Cardiomyopathy Questionnaire improvement by >10)

CONTACTS AND LOCATIONS:
Overall Officials: Vinny Podichetty, Study Director — VDyne, Inc.
Locations (21):
- Australia (5):
  - St. Vincent Hospital, Sydney, New South Wales
  - Flinders Medical Centre, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - The Prince Charles Hospital, Brisbane
  - Monash Heart, Melbourne
- Austria (2):
  - Johannes Kepler University Linz - JKU, Linz
  - Universitätsklinik für Herzchirurgie Medizinische Universität Wien, Vienna
- AZ Sint Jan Hospital, Bruges, Belgium
- Nemocnice AGEL Podlesi Trinec, Třinec, Czechia
- University Hospital of Copenhagen, Copenhagen, Denmark
- Germany (4):
  - Herz & Diabeteszentrum Nordrhein Westfalen, Bad Oeynhausen
  - Vivantes Klinik Am Urban, Berlin
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsmedizin Rostock, Rostock
- St Antonius Hospital, Nieuwegein, Netherlands
- Waikato Hospital, Hamilton, Hamilton, New Zealand
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico San Carlos, Madrid
- Lund University Skåne University Hospital, Lund, Sweden
- United Kingdom (2):
  - Royal Sussex Hospital, Brighton, Sussex
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.